CLINICAL TRIAL: NCT06172296
Title: A Phase 3 Study of Dinutuximab Added to Intensive Multimodal Therapy for Children With Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Dinutuximab With Chemotherapy, Surgery and Stem Cell Transplantation for the Treatment of Children With Newly Diagnosed High Risk Neuroblastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-08530; NCI-2023-08530 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL2131 (Other: Children's Oncology Group); ANBL2131 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2023-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Ganglioneuroblastoma, Nodular; Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — Specimen Handling; Biopsy; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; dinutuximab; Doxorubicin; Etoposide; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Irinotecan; Isotretinoin; Leukapheresis; Magnetic Resonance Spectroscopy; Melphalan; Radiotherapy; Radiation; Nuclear Medicine Department, Hospital; Temozolomide; Thiotepa; Topotecan; Transurethral Resection of Bladder; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (SOC treatment) (Active Comparator): See detailed description
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dinutuximab; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Etoposide; Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan; Procedure: Hematopoietic Cell Transplantation; Drug: Irinotecan; Drug: Isotretinoin; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Radiation: Radiation Therapy; Procedure: Radionuclide Imaging; Other: Survey Administration; Drug: Temozolomide; Drug: Thiotepa; Drug: Topotecan; Procedure: Tumor Resection; Drug: Vincristine
- Arm B (Dinutuximab in induction) (Experimental): See detailed description
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dinutuximab; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Etoposide; Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan; Procedure: Hematopoietic Cell Transplantation; Drug: Irinotecan; Drug: Isotretinoin; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Radiation: Radiation Therapy; Procedure: Radionuclide Imaging; Other: Survey Administration; Drug: Temozolomide; Drug: Thiotepa; Drug: Topotecan; Procedure: Tumor Resection; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Procedure: FDG-Positron Emission Tomography and Computed Tomography Scan — Undergo FDG PET
  Other Names: FDG PET/CT
Procedure: Hematopoietic Cell Transplantation — Undergo stem cell infusion
  Other Names: HCT; Hematopoietic Stem Cell Infusion; HEMATOPOIETIC STEM CELL TRANSPLANT; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; Stem Cell Transplantation, NOS
Drug: Irinotecan — Given IV
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Procedure: Leukapheresis — Undergo apheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Radionuclide Imaging — Undergo I-MIBG scan
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Other: Survey Administration — Ancillary studies
Drug: Temozolomide — Given PO or via NG or G tube
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
Procedure: Tumor Resection — Undergo tumor resection surgery
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase III trial tests how well the addition of dinutuximab to Induction chemotherapy along with standard of care surgical resection of the primary tumor, radiation, stem cell transplantation, and immunotherapy works for treating children with newly diagnosed high-risk neuroblastoma. Dinutuximab is a monoclonal antibody that binds to a molecule called GD2, which is found on the surface of neuroblastoma cells, but is not present on many healthy or normal cells in the body. When dinutuximab binds to the neuroblastoma cells, it helps signal the immune system to kill the tumor cells. This helps the cells of the immune system kill the cancer cells, this is a type of immunotherapy. When chemotherapy and immunotherapy are given together, during the same treatment cycle, it is called chemoimmunotherapy. This clinical trial randomly assigns patients to receive either standard chemotherapy and surgery or chemoimmunotherapy (chemotherapy plus dinutuximab) and surgery during Induction therapy. Chemotherapy drugs administered during Induction include, cyclophosphamide, topotecan, cisplatin, etoposide, vincristine, and doxorubicin. These drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing or by stopping them from spreading. Upon completion of 5 cycles of Induction therapy, a disease evaluation is completed to determine how well the treatment worked. If the tumor responds to therapy, patients receive a tandem transplantation with stem cell rescue. If the tumor has little improvement or worsens, patients receive chemoimmunotherapy on Extended Induction. During Extended Induction, dinutuximab is given with irinotecan, temozolomide. Patients with a good response to therapy move on to Consolidation therapy, when very high doses of chemotherapy are given at two separate points to kill any remaining cancer cells. Following, transplant, radiation therapy is given to the site where the cancer originated (primary site) and to any other areas that are still active at the end of Induction. The final stage of therapy is Post-Consolidation. During Post-Consolidation, dinutuximab is given with isotretinoin, with the goal of maintaining the response achieved with the previous therapy. Adding dinutuximab to Induction chemotherapy along with standard of care surgical resection of the primary tumor, radiation, stem cell transplantation, and immunotherapy may be better at treating children with newly diagnosed high-risk neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the event-free survival (EFS) of patients with newly diagnosed high-risk neuroblastoma assigned to early chemoimmunotherapy during Induction differs from that of patients who are not assigned to treatment that includes early chemoimmunotherapy.

SECONDARY OBJECTIVES:

I. To determine if early chemoimmunotherapy during Induction therapy improves end of Induction (EOI) response rates and overall survival (OS) for patients with newly diagnosed high-risk neuroblastoma.

II. To determine response rates, EFS, and OS following an Extended Induction regimen with chemoimmunotherapy in patients with progressive disease or a poor response to Induction therapy.

III. To compare the toxicities experienced by patients treated with chemoimmunotherapy during Induction versus those experienced by patients treated with standard Induction and to describe toxicities experienced during Extended Induction.

IV. To determine GD2 expression on tumor tissue and tumor cells in bone marrow and assess for associations with response and outcome.

EXPLORATORY OBJECTIVES:

I. To describe the association between tumor and host factors and outcomes in patients receiving protocol therapy.

II. To evaluate circulating biomarkers and markers of minimal residual disease at baseline and during therapy, and assess for associations with response and outcome.

III. To compare patterns of failure between patients treated with and without dinutuximab during induction.

IV. To determine the effect of telomere maintenance mechanisms on end of Induction response rates, EFS, and OS.

V. To explore the impact of high-risk neuroblastoma (HRNBL) and its therapy, including the addition of dinutuximab to Induction chemotherapy, on functional and quality of life outcomes in patients with HRNBL, as measured by caregiver (parent/legal guardian) and patient questionnaires.

VI. To describe the adequacy of diagnostic biopsy specimens, including those obtained by percutaneous core needle biopsy.

VII. To explore the associations between family-reported adverse social determinants of health and both clinical outcomes and biology.

VIII. To develop and validate deep learning predictors of Induction response based on diagnostic MIBG scans. (Imaging Objective) IX. To compare institutional versus central determination of overall response, individual response components (primary tumor, soft tissue and bone metastatic disease, and bone marrow metastatic disease), and poor end of induction response (PEIR) and good end of induction response (GEIR) determination. (Imaging Objective) X. To describe late toxicities (including impaired organ function, neuropsychiatric toxicity, and incidence of secondary malignancy) in patients treated with dinutuximab during Induction or Extended Induction to late toxicities in patients who have not received dinutuximab during these phases of therapy.

XI. To evaluate whether reduced dose radiotherapy to the primary site clinical target volume (CTV) in patients with complete response of the primary site at EOI results in comparable local control relative to historical cohorts.

XII. To compare post-transplant complications between treatment arms, and assess for associations with outcome.

XIII. To assess for associations between EOI response (including good end of Induction response [GEIR] and poor end of Induction response [PEIR]) and individual response components (primary tumor, soft tissue and bone metastatic disease, and bone marrow metastatic disease) with outcome (EFS and OS).

XIV. To describe and compare the changes in image-defined risk factors (IDRFs) between patients treated with and without dinutuximab during Induction and associate with surgical outcomes and local failure rates following primary tumor resection.

XV. To bank serial samples of blood, bone marrow, and tumor tissue for future research.

OUTLINE: Patients receive Induction cycle 1 and are then randomized to 1 of 2 treatment arms.

INDUCTION CYCLE 1: Patients receive cyclophosphamide intravenously (IV) over 30 minutes and topotecan IV over 30 minutes on days 1-5 in the absence of unacceptable toxicity.

ARM A:

INDUCTION CYCLES 2-5: Patients receive cyclophosphamide IV over 30 minutes and topotecan IV over 30 minutes on days 1-5 of cycle 2 in the absence of unacceptable toxicity. Patients then undergo stem cell harvest via apheresis. Patients then receive cisplatin IV over 4 hours and etoposide IV over 2 hours on days 1-3 of cycles 3 and 5, and vincristine IV on day 1, doxorubicin IV over 15 minutes, and cyclophosphamide IV over 1 hour on days 1-2 of cycle 4 in the absence of unacceptable toxicity. Patients undergo primary tumor resection after Induction cycle 4 or 5. Following Induction cycle 5, patients undergo testing to determine response to Induction therapy. Patients with a good tumor response proceed to Consolidation, while patients with a poor tumor response proceed to Extended Induction.

EXTENDED INDUCTION: Patients with a poor tumor response or progression during Induction receive temozolomide orally (PO), via nasogastric tube (NG), or via gastric tube (G-tube) on days 1-5, irinotecan IV over 90 minutes on days 1-5, and dinutuximab IV over 10 hours. Treatment repeats every 21 days for up to a maximum of 6 cycles in the absence of disease progression or unacceptable toxicity. If at any time during Extended Induction testing shows a good tumor response, patients proceed to Consolidation. If after 6 cycles of Extended Induction or if at any time progression is noted, patients are removed from the study.

CONSOLIDATION: Patients undergo two autologous hematopoietic stem cell transplantations (HSCTs) during Consolidation. Patients receive thiotepa IV over 2 hours on days -7 to -5 and cyclophosphamide IV over 1 hour on days -5 to -2 during HSCT 1. Patients then receive stem cell infusion IV on day 0. Between 6 and 10 weeks after stem cell infusion, patients receive melphalan IV over 30 minutes on days -7 to -5, etoposide IV over 24 hours on days -7 to -4, and carboplatin over 24 hours on days -7 to -4 during HSCT 2. Patients receive stem cell infusion IV on day 0. Between day +42 and day +80 after HSCT 2. Patients receive radiation daily for 12 treatments in the absence of disease progression or unacceptable toxicity.

POST CONSOLIDATION: Patients receive dinutuximab IV over 10 hours on days 4-7 and isotretinoin PO twice daily (BID) on days 11-24 of cycles 1-5. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive isotretinoin PO BID on days 15-28 for 1 additional cycle, cycle 6.

Patients undergo blood and urine sample collection, echocardiogram (ECHO) or multigated acquisition scan (MUGA), bone marrow aspiration and/or biopsy, computed tomography (CT) scan, magnetic resonance imaging (MRI), iodine-123 meta-iodobenzylguanidine (I-MIBG) scan and possible fluorodeoxyglucose position emission tomography (FDG-PET) scan throughout the study.

ARM B:

INDUCTION CYCLES 2-5: Patients receive cyclophosphamide IV over 30 minutes, topotecan IV over 30 minutes on days 1-5, and dinutuximab IV over 10 hours on days 2-5 of cycle 2 in the absence of unacceptable toxicity. Patients then undergo stem cell harvest via apheresis. Patients receive cisplatin IV over 4 hours and etoposide IV over 2 hours on days 1-3 and dinutuximab IV over 10 hours on days 2-5 of cycles 3 and 5, and vincristine IV on day 1, doxorubicin IV over 15 minutes, and cyclophosphamide IV over 1 hour on days 1-2, and dinutuximab IV over 10 hours on days 2-5 of cycle 4 in the absence of unacceptable toxicity. Patients undergo primary tumor resection after Induction cycle 4 or 5. Following Induction cycle 5, patients undergo testing to determine response to Induction therapy. Patients with a good tumor response proceed to Consolidation, while patients with a poor tumor response proceed to Extended Induction.

EXTENDED INDUCTION: Patients with a poor tumor response or progression during Induction receive temozolomide PO, via NG tube, or via G-tube on days 1-5, irinotecan IV over 90 minutes on days 1-5, and dinutuximab IV over 10 hours. Treatment repeats every 21 days for up to a maximum of 6 cycles in the absence of disease progression or unacceptable toxicity. If at any time during Extended Induction testing shows a good tumor response, patients proceed to Consolidation. If after 6 cycles of Extended Induction or if at any time progression is noted, patients are removed from the study.

CONSOLIDATION: Patients undergo two autologous HSCTs during Consolidation. Patients receive thiotepa IV over 2 hours on days -7 to -5 and cyclophosphamide IV over 1 hour on days -5 to -2 during HSCT 1. Patients then receive stem cell infusion IV on day 0. Between 6 and 10 weeks after stem cell infusion patients receive melphalan IV over 30 minutes on days -7 to -5, etoposide IV over 24 hours on days -7 to -4, and carboplatin over 24 hours on days -7 to -4 during HSCT 2. Patients receive stem cell infusion IV on day 0. Between day +42 and day +80 after HSCT 2, patients receive radiation daily for 12 treatments in the absence of disease progression or unacceptable toxicity.

POST CONSOLIDATION: Patients receive dinutuximab IV over 10 hours on days 4-7 and isotretinoin PO BID on days 11-24 of cycles 1-5. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive isotretinoin PO BID on days 15-28 for 1 additional cycle, cycle 6.

Patients undergo blood and urine sample collection, ECHO or MUGA, bone marrow aspiration and/or biopsy, CT scan, MRI, I-MIBG scan and possible FDG-PET scan throughout the study.

After completion of study treatment, patients are followed up at 3, 6, 9,12, 15, 18, 24, 30, 36, 42, 48, 54, and 60 months and then periodically for up to 10 years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on APEC14B1 and have consented to testing through the Molecular Characterization Initiative (MCI), prior to enrollment on ANBL2131
* ≤ 30 years at the time of initial diagnosis with high-risk disease
* * Must have a diagnosis of neuroblastoma (NBL) or ganglioneuroblastoma (nodular) verified by tumor pathology analysis or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamines

  * Newly diagnosed, high risk neuroblastoma (HRNBL) defined as one of the following:

    * Any age with International Neuroblastoma Risk Group (INRG) Stage L2, MS, or M and MYCN amplification
    * Age ≥ 547 days and INRG stage M regardless of biologic features (clinical MYCN testing not required prior to enrollment)
    * Any age initially diagnosed with INRG Stage L1 MYCN amplified NBL who have progressed to stage M without systemic chemotherapy
    * Age ≥ 547 days of age initially diagnosed with INRG Stage L1, L2, or MS who have progressed to stage M without systemic chemotherapy (clinical MYCN testing not required prior to enrollment)
* Patients must have a body surface area (BSA) ≥ 0.25 m^2
* No prior anti-cancer therapy except as outlined below:

  * Patients initially recognized to have high-risk disease treated with topotecan/cyclophosphamide initiated on an emergent basis and within allowed timing, and with consent
  * Patients observed or treated with a single cycle of chemotherapy per a low or intermediate risk neuroblastoma regimen (e.g., as per ANBL0531, ANBL1232 or similar) for what initially appeared to be non-high-risk disease but subsequently found to meet the criteria
  * Patients who received localized emergency radiation to sites of life threatening or function-threatening disease prior to or immediately after establishment of the definitive diagnosis
* Human immunodeficiency virus (HIV) -infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* A serum creatinine based on age/sex as follows:

  * 1 month to < 6 months: Male 0.4 mg/dL and female 0.4mg/dL
  * 6 months to < 1 year: Male 0.5 mg/dL and female 0.5 mg/dL
  * 1 to < 2 years: Male 0.6 mg/dL and female 0.6 mg/dL
  * 2 to < 6 years: Male 0.8 mg/dL and female 0.8 mg/dL
  * 6 to < 10 years: Male 1 mg/dL and female 1 mg/dL
  * 10 to < 13 years: Male 1.2 mg/dL and female 1.2 mg/dL
  * 13 to < 16 years: Male 1.5 mg/dL and female 1.4 mg/dL
  * ≥ 16 years: Male 1.7 mg/dL and female 1.4 mg/dL

    * The threshold creatinine values were derived from the Schwartz formula for estimating glomerular filtration rate (GFR) utilizing child length and stature data published by the Centers for Disease Control (CDC)
  * or a 24-hour urine creatinine clearance ≥ 70 mL/min/1.73 m^2 or
  * or a GFR ≥ 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method or direct small molecule clearance method (iothalamate or other molecule per institutional standard)

    * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
* Serum glutamic pyruvic transaminase (SGPT) (Alanine aminotransferase [ALT]) ≤ 10 x ULN*

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* * Shortening fraction of ≥ 27% by echocardiogram, or

  * Ejection fraction of ≥ 50% by echocardiogram or radionuclide angiogram
* Ability to tolerate Peripheral Blood Stem Cell (PBSC) collection:

No known contraindication to PBSC collection. Examples of contraindications might be a weight or size less than the collecting institution finds feasible, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure

Exclusion Criteria:

* Patients who are 365-546 days of age with INRG Stage M and MYCN non-amplified NBL, irrespective of additional biologic features
* Patients ≥ 547 days of age with INRG Stage L2, MYCN non-amplified NBL, regardless of additional biologic features
* Patients with known bone marrow failure syndromes
* Patients on chronic immunosuppressive medications (e.g., tacrolimus, cyclosporine, corticosteroids) for reasons other than prevention/treatment of allergic reactions and adrenal replacement therapy are not eligible. Topical and inhaled corticosteroids are acceptable
* Patients with a primary immunodeficiency syndrome who require ongoing immune globulin replacement therapy
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required prior to enrollment for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, food and drug administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 478 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | Up to 3 years
  EFS time is calculated from time of randomization to Arms A or B to first episode of disease relapse or progression, second malignancy, or death, or until last contact if no event has occurred.

SECONDARY OUTCOMES:
End of Induction (EOI) response rate | From randomization to end of extended Induction, up to 12 months
  The response rate will be calculated among all evaluable patients at end of Induction. Responders are defined as patients who achieve a >= partial response per the revised 2017 International Neuroblastoma Response Criteria (INRC)
Overall survival (OS) | Up to 3 years
  OS time is calculated from time of randomization to Arms A or B until death, or until last contact if patient is alive.
Incidence of adverse events | Up to 2 years
  The proportion of patients with at least one grade 3 or higher non-hematologic toxicity or grade 4 or higher hematologic toxicity during protocol therapy, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, will be reported.
GD2 expression | Up to 12 months
  Dinutuximab binding to pre-therapy patient tumor samples will be measured and categorized as high or low.

OTHER OUTCOMES:
Association between tumor and host factors and outcomes | Up to 10 years
  A series of univariate and multivariate Cox proportional hazards (for EFS and OS) and logistic regression (for responders vs. non-responders) models will be fit for patients in Arms A and B to evaluate the relationship between tumor and host factors (including tumor ALK and other somatic mutations, copy-number aberrations, gene fusions, gene expression, and pathogenic germline variants) and chemo-immunotherapy during Induction with outcome.
Circulating biomarkers and markers of minimal residual disease | Up to 10 years
  Will be assessed by comparing the proportion of patients with detectable vs. non-detectable tumor markers (including circulating tumor deoxyribonucleic acid, circulating free DNA, circulating tumor cells, and immune function profiling) between Arms A and B during and after induction and post-consolidation therapy using chi-squared tests at each individual time point, and Cochran's Q across time points to determine if there is a consistent difference in proportions between arms across time. In addition, the tumor markers will be analyzed as continuous variables using longitudinal data analysis methodology such as mixed effects models or generalized estimating equations as appropriate.
Patterns of failure | Up to 10 years
  The impact of early or late chemoimmunotherapy during Induction on the probability of the involvement of a specific disease site at first relapse will be evaluated using Fisher's exact test.
Effect of telomere maintenance mechanisms | Up to 10 years
  A series of univariate and multivariate Cox proportional hazards (for EFS and OS) and logistic regression (for responders vs. non-responders) models will be fit for patients in arms A and B to evaluate the relationship between telomere maintenance mechanism and chemoimmunotherapy during Induction with outcome. Patients will be classified into 3 groups by telomere maintenance mechanism (TMM) based on messenger ribonucleic acid expression of TERT and analysis of telomeric DNA C-circles: telomerase (TERT) positive, alternative of lengthening of telomeres (ALT) positive, or no identified TMM.
Functional and quality of life outcomes | At serial time points during Induction, Extended Induction, Post-Consolidation, and at the end of therapy
  Will descriptively summarize and compare the total Memorial Symptom Assessment Scale scores, total sub-domain scores, and individual symptom scores between patients randomized to receive dinutuximab during Induction (Arm B) to those of patients randomized to standard Induction (Arm A).
Adequacy of diagnostic biopsy specimens | At time of tissue collection
  Will be evaluated by descriptively comparing the successful delineation of histologic classification, MYCN amplification status, and ALK status via the traditional method of obtaining tissue for diagnosis, open surgical biopsy, versus the less invasive percutaneous core needle biopsy.
Associations between family-reported adverse social determinants of health and both clinical outcomes and biology | Up to 10 years
  Kaplan-Meier curves of EFS and OS will be generated and used to calculate 3-year EFS and OS estimates. Associations between social determinants of health (SDOH) and survival outcomes and time to receipt of dinutuximab will be evaluated with univariate and multivariate Cox proportional hazard models. Log-binomial regression will be used to estimate risk ratios and 95% CI for the occurrence of dinutuximab consent to randomization and therapy receipt by SDOH exposure. Effect modification of outcomes as a function of poverty, stratified by race/ethnicity, will be explored.
Develop and validate deep learning predictors of Induction response (imaging objective) | At diagnosis, EOI, during Extended Induction, and end of Extended Induction
  Scans will be given as input to a convolutional neural network trained to predict EOI response.
Compare institutional versus central determination of overall response, individual response components, and PEIR and GEIR determination (imaging objective) | Up to 10 years
  Will be assessed by calculating the percentage of patients receiving the same EOI institutional and centrally reviewed determination of overall response, individual response components (primary tumor, soft tissue and bone metastatic disease, and bone marrow metastatic disease), and PEIR and GEIR. In addition, Cohen's kappa will be calculated to evaluate the concordance in each of these response measures.
Incidence of late toxicities | Up to 10 years
  Will be addressed by calculating the proportion of treated patients with each late effect, including but not limited to impaired organ function, neuropsychiatric toxicity, and secondary malignancy. A 95% confidence interval will be placed on each proportion.
Reduced dose radiotherapy to the primary site clinical target volume (CTV) in patients with complete response of the primary site at EOI results in comparable local control relative to historical cohorts | Up to 10 years
  The cumulative incidence of local progression (CILP) in patients with complete response of the primary site at EOI and GEIR on this study will be compared to the CILP rate of 11.2±1.8% observed on ANBL0532 using Gray's test.
Post-transplant complications | Up to 100 days post-transplant
  Will be evaluated by calculating the incidence of endothelial injury complications and non-relapse mortality within 100 days of transplant, transplant-associated thrombotic microangiopathy (TA-TMA), severe TA-TMA, and sinusoidal obstruction syndrome (SOS) on Arms A and B and comparing between arms with a chi-squared test. The impact of TA-TMA occurrence on the timing or exclusion of subsequent therapy and interventions utilized to treat the TA-TMA, and associations with outcomes (EFS and OS) will be assessed.
Associations between end of induction (EOI) response and individual response components | Up to 10 years
  Log-rank tests will be used to explore the association between EOI response (using both the revised INRC and GEIR/PEIR classification) and individual response components (primary tumor, soft tissue and bone metastatic disease, and bone marrow metastatic disease) with outcome (EFS and OS).
Changes in image-defined risk factors (IDRF) | Up to 10 years
  The proportion of patients in the analytic cohort for whom each particular IDRF and also the presence of any IDRF is absent prior to surgical resection will be computed. McNemar's test for paired observations will be applied to determine whether there is a difference in the proportion of each IDRF and any IDRF present before and after initial therapy, and conditional logistic regression will be used to compare between treatment arms A and B. The IDRF status after initial therapy and whether there has been a change from diagnosis will be associated with surgical outcome (complete vs. incomplete resection, presence or absence of surgical complications) using chi-squared tests, and compared between treatment arms A and B with the Cochran-Mantel-Haenszel test. The association of IDRF status with presence or absence of local failure after primary tumor resection will also be evaluated using a chi-squared test, and compared between treatment arms A and B with the Cochran-Mantel-Haenszel.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Federico, Principal Investigator — Children's Oncology Group
Locations (174):
- United States (153):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Starship Children's Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm